CLINICAL TRIAL: NCT01713348
Title: Sensor and Software Use for Improved Glucose Control in MDI Managed Diabetes
Acronym: SIGN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ADC-PMR-APO-12015
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus
Keywords: CGM; MDI
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGM - intervention arm (Experimental): Following a 14 day masked (baseline) period using the FreeStyle Navigator subjects will wear an unmasked FreeStyle Navigator with the glucose alarms switched off.
  Interventions: Device: FreeStyle Navigator
- SMBG - Control arm (Active Comparator): Following a 14 day masked ( baseline) period using the FreeStyle Navigator subjects will manage their blood glucose with a standard SMBG and use a FreeStyle Navigator masked for a 14 day period at the end of the study.
  Interventions: Device: Standard SMBG

INTERVENTIONS:
Device: FreeStyle Navigator — Masked CGM day 1 to 15, unmasked CGM days 15 to 100
  Arms: CGM - intervention arm
Device: Standard SMBG — Masked CGM days 1 to 15, standard SMBG days 15 to 86, masked CGM day 86 to 100
  Arms: SMBG - Control arm

SUMMARY:
To understand if Multiple Daily Injections (MDI) managed subjects can improve glycaemic control by;

1. regularly checking and understanding Continuous Glucose data & trend arrows at times other than the standard pre-meal bolus calculation test times and
2. review of their glucose profiles (inc. hypoglycaemic risks) with their Health Care Professional (HCP) and adjusting behaviours & therapy from interpretation of the Continuous Glucose profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Type 1 diabetes on MDI with bolus injections for >6 months prior to study enrolment or Type 2 diabetes treated with 2 or more insulin injections daily.
* In the investigator's opinion, thought technically capable of using FreeStyle Navigator GM System device.
* HbA1c between 7.5 and 12.0% (58 to 108 mmol/mol) for previous test obtained within 6 months prior to point of enrolment

Exclusion Criteria:

* Concomitant disease or condition that may compromise patient safety, including unstable coronary heart disease, cystic fibrosis, serious psychiatric disorder, or any uncontrolled chronic medical condition
* Female subject is pregnant or planning to become pregnant within the planned study duration. Subjects who become pregnant during the study will be discontinued from the study.
* Currently using / has previously used a Continuous Glucose Monitoring System within the last 6 months.
* Currently using Continuous Subcutaneous Insulin Infusion (CSII)
* Currently using basal/long acting insulin only.
* Participating in another study of a glucose monitoring device / drug that could affect glucose measurements / management
* Known allergy to medical grade adhesives
* In the investigators opinion is unsuitable to participate due to any other cause/reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Ajjan, Principal Investigator — St James Hospital, Leeds
Locations (9):
- United Kingdom (9):
  - Ayr Hospital, Ayr, Ayrshire
  - Tameside Hospital NHS Foundation Trust, Ashton-under-Lyne
  - Royal United Hospital, Bath
  - Birmingham Heartlands Hospital, Diabetes Clinic, City and Borough of Birmingham
  - University Hospital of North Durham, Durham
  - Ipswich Hospital NHS Trust, Ipswich
  - St James Hospital,, Leeds
  - Rotherham General Hospital, Rotherham
  - Diabetes Centre, New Cross Hospital,, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 105 subjects consented and enrolled into the study. Eighteen of these withdrew before randomisation or failed screening. Eighty-seven (87) subjects were randomised and 79 completed the study.
Groups:
- CGM - Intervention Arm - Type 1 Diabetes; CGM - Intervention Arm - Type 2 Diabetes: Following a 14 day masked (baseline) period using the FreeStyle Navigator subjects will wear an unmasked FreeStyle Navigator with the glucose alarms switched off.
  FreeStyle Navigator: Masked CGM day 1 to 15, unmasked CGM days 15 to 100
- SMBG - Control Arm - Type 1 Diabetes; SMBG - Control Arm - Type 2 Diabetes: Following a 14 day masked ( baseline) period using the FreeStyle Navigator subjects will manage their blood glucose with a standard SMBG and use a FreeStyle Navigator masked for a 14 day period at the end of the study.
  Standard SMBG: Masked CGM days 1 to 15, standard SMBG days 15 to 86, masked CGM day 86 to 100
Period: Overall Study
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Started | 29 | 13 | 30 | 15
Completed | 25 | 11 | 28 | 15
Not Completed | 4 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes | Total
Number analyzed (Participants) | 29 | 13 | 30 | 15 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.5) | 43.7 (9.9) | 57.8 (8.8) | 55.5 (10.9) | 49.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 11 | 4 | 36
  Male | 15 | 6 | 19 | 11 | 51
Region of Enrollment [Number; unit: participants]
  United Kingdom | 29 | 13 | 30 | 15 | 87
Baseline HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 76.4 (14.1) | 74.8 (13.9) | 76.5 (15.0) | 77.4 (13.7) | 76.4 (14.1)
Baseline HbA1c [Mean (Standard Deviation); unit: %] | 9.2 (1.3) | 9.0 (1.3) | 9.2 (1.4) | 9.2 (1.3) | 9.1 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Time in Range
Description: Intervention arm: within subject difference in time in range (70-180 mg/dL, 3.9 to 10.0 mmol/L) in final 15 days compared to baseline phase assessed separately for Type 1 and Type 2 Diabetes.
Time Frame: Day 86 to 100 compared to Day 1 to 15
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Number analyzed (Participants) | 29 | 11 | 28 | 15
hours per day
  Baseline | 10.9 (3.0) | 11.5 (4.6) | 13.3 (5.2) | 12.3 (7.0)
  Final | 10.8 (3.9) | 11.5 (4.2) | 14.7 (5.8) | 13.3 (5.5)
Statistical Analysis 1: Comparison: CGM - Intervention Arm - Type 1 Diabetes; Test type: Superiority or Other; p = 0.9345, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.29 to 1.19], Standard Deviation 3.3
Statistical Analysis 2: Comparison: CGM - Intervention Arm - Type 2 Diabetes; Difference in time in range (70-180 mg/dL, 3.9 to 10.0 mmol/L) intervention arm compared to control arm; Test type: Superiority or Other; p = 0.0427, t-test, 2 sided; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [0.05 to 2.73], Standard Deviation 3.5

2. Secondary Outcome: Time in Range
Description: Difference in time in range (70-180 mg/dL, 3.9 to 10.0 mmol/L) intervention arm compared to control arm.
Time Frame: Days 86 to 100 intervention arm compared to control arm
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Number analyzed (Participants) | 29 | 11 | 28 | 15
hours per day
  Baseline | 10.9 (3.0) | 11.5 (4.6) | 13.3 (5.2) | 12.3 (7.0)
  Final | 10.8 (3.9) | 11.5 (4.2) | 14.7 (5.8) | 13.3 (5.5)
Statistical Analysis 1: Comparison: CGM - Intervention Arm - Type 1 Diabetes vs SMBG - Control Arm - Type 1 Diabetes; Test type: Superiority or Other; p = 0.8367, ANCOVA; Performed for each type of Diabetes and adjusted for baseline Time in Range; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-2.65 to 2.16], Standard Deviation 1.18
Statistical Analysis 2: Comparison: CGM - Intervention Arm - Type 2 Diabetes vs SMBG - Control Arm - Type 2 Diabetes; Test type: Superiority or Other; p = 0.7969, ANCOVA; Performed for each type of Diabetes and adjusted for baseline Time in Range; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-1.86 to 2.40], Standard Deviation 1.05

3. Secondary Outcome: Glucose Standard Deviation (SD)
Time Frame: Day 86 to 100 compared to day 1 to 15
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Number analyzed (Participants) | 29 | 11 | 28 | 15
mmol/L
  Baseline | 4.0 (0.8) | 3.7 (0.8) | 3.0 (0.7) | 3.1 (1.0)
  Final | 3.8 (0.7) | 3.8 (0.6) | 2.8 (0.7) | 3.0 (0.6)
Statistical Analysis 1: Comparison: CGM - Intervention Arm - Type 1 Diabetes; Test type: Superiority or Other; p = 0.0352, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.51 to -0.02], Standard Deviation 0.6
Statistical Analysis 2: Comparison: CGM - Intervention Arm - Type 2 Diabetes; Test type: Superiority or Other; p = 0.0506, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.54 to 0.00], Standard Deviation 0.7

4. Secondary Outcome: HbA1c (mmol/Mol)
Time Frame: Day 100 compared to day 1
Population: Analysis performed according to the intention-to-treat principle. Analysis in the Type 1 population is after removal of 1 outlier.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Number analyzed (Participants) | 28 | 13 | 30 | 15
mmol/mol
  Baseline | 75 (10) | 75 (14) | 77 (15) | 77 (14)
  Final | 72 (8) | 74 (14) | 67 (13) | 72 (9)
Statistical Analysis 1: Comparison: CGM - Intervention Arm - Type 1 Diabetes; Test type: Superiority or Other; p = 0.0580, t-test, 2 sided; Mean Difference (Final Values) = -3, 95% CI 2-sided [-6.4 to 0.1], Standard Deviation 8
Statistical Analysis 2: Comparison: CGM - Intervention Arm - Type 2 Diabetes; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided; Mean Difference (Final Values) = -9, 95% CI 2-sided [-13.6 to -4.9], Standard Deviation 12

5. Secondary Outcome: HbA1c
Time Frame: Day 100 compared to day 1
Population: Analysis performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Number analyzed (Participants) | 28 | 13 | 30 | 15
Percent
  Baseline | 9.0 (0.9) | 9.0 (1.3) | 9.2 (1.4) | 9.2 (1.3)
  Final | 8.7 (0.7) | 8.9 (1.3) | 8.3 (1.2) | 8.8 (0.8)
Statistical Analysis 1: Comparison: CGM - Intervention Arm - Type 1 Diabetes; Test type: Superiority or Other; p = 0.0580, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.59 to 0.01], Standard Deviation 0.8
Statistical Analysis 2: Comparison: CGM - Intervention Arm - Type 2 Diabetes; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.24 to -0.45], Standard Deviation 1.1

ADVERSE EVENTS:
Time Frame: Adverse events collected from enrollment to completion by last subject (8 months)
Description: In addition to the adverse events listed below, one subject who withdrew from the study before randomisation reported Menieres disease.
Arm/Group | CGM - Intervention Arm - Type 1 Diabetes | SMBG - Control Arm - Type 1 Diabetes | CGM - Intervention Arm - Type 2 Diabetes | SMBG - Control Arm - Type 2 Diabetes
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/13 | 0/30 | 1/15
Other Adverse Events (participants affected / at risk) | 13/29 | 7/13 | 17/30 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM - Intervention Arm - Type 1 Diabetes (N=29) | SMBG - Control Arm - Type 1 Diabetes (N=13) | CGM - Intervention Arm - Type 2 Diabetes (N=30) | SMBG - Control Arm - Type 2 Diabetes (N=15)
Severe hypoglycaemia (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Not device or study related.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not device or study related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM - Intervention Arm - Type 1 Diabetes (N=29) | SMBG - Control Arm - Type 1 Diabetes (N=13) | CGM - Intervention Arm - Type 2 Diabetes (N=30) | SMBG - Control Arm - Type 2 Diabetes (N=15)
Hypoglycaemia (Endocrine disorders) | 3 (10) | 1 (4) | 2 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sensor tip (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cold (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 4 (6) | 8 (11) | 3 (3)
Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 6 (9)
Sickness (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Infection - general (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Allergic reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - renal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dental (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days